CLINICAL TRIAL: NCT02266277
Title: System Alignment for VaccinE Delivery (SAVED): Improving Rates of Influenza and Pneumococcal Vaccination Through Patient Outreach, Improved Medical Record Accuracy and Targeted Physician Alerts.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Massachusetts, Worcester (Other)
Collaborators: Reliant Medical Group (Other); Pfizer (Industry)
Responsible Party: Principal Investigator, Sarah Cutrona, Assistant Professor of Medicine, University of Massachusetts, Worcester
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Health Services Research
Other Study IDs: 9713747; H00006928 (Other: University of Massachusetts Medical School IRB)
Record Dates: First submitted 2014-10-10; First posted 2014-10-17 (Estimated); Results first posted 2017-03-28 (Actual); Last update posted 2017-05-31 (Actual); Status verified 2017-05

CONDITIONS: Influenza; Infections, Pneumococcal
Keywords: electronic health record, utilization; randomized controlled trial; pragmatic clinical trial; influenza, prevention and control; pneumococcal vaccines; qualitative research
MeSH Terms: conditions — Influenza, Human; Pneumococcal Infections; Patient Acceptance of Health Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- Arm 1: E-portal message with IVR call (Active Comparator): Patients identified as e-portal users will receive an e-portal message with IVR call
  Interventions: Other: Arm 1: E-portal message with IVR call
- Arm 2: E-portal message with no IVR call (Active Comparator): Patients identified as e-portal users will receive an e-portal message only
  Interventions: Other: Arm 2: E-portal message with no IVR call
- Arm 3: No e-portal message with IVR call (Active Comparator): Patients identified as e-portal users will receive an IVR call only
  Interventions: Other: Arm 3: No e-portal message with IVR call
- Arm 4: No E-portal message with no IVR call (No Intervention): Patients identified as e-portal users will receive neither an e-portal message nor an IVR call
- Arm 5: IVR call (Active Comparator): Patients identified as non e-portal users will receive an IVR call only
  Interventions: Other: Arm 5: IVR call
- Arm 6: No IVR call (No Intervention): Patients identified as non e-portal users will not receive any outreach

INTERVENTIONS:
Other: Arm 1: E-portal message with IVR call — Active electronic patient portal users will be randomized to receive an e-portal message and IVR calls. Both methods of outreach will provide patients with educational information about influenza vaccination, notify patients of local flu clinic schedules and elicit patient response to vaccination status and barriers.
  Arms: Arm 1: E-portal message with IVR call
Other: Arm 2: E-portal message with no IVR call — Active electronic patient portal users will be randomized to receive only an e-portal message. The e-portal message will provide patients with educational information about influenza vaccination, notification of local flu clinic schedules and elicit patient response to vaccination status and barriers.
  Arms: Arm 2: E-portal message with no IVR call
Other: Arm 3: No e-portal message with IVR call — Active electronic patient portal users will be randomized to receive an IVR call. The IVR call will provide patients with educational information about influenza vaccination, notification of local flu clinic schedules and elicit patient response to vaccination status and barriers.
  Arms: Arm 3: No e-portal message with IVR call
Other: Arm 5: IVR call — Non electronic patient portal users will be randomized to receive an IVR call with educational information about influenza vaccines, notification of local flu clinic schedules and elicit patient response to vaccination status and barriers.
  Arms: Arm 5: IVR call

SUMMARY:
The goal of this research study is to improve rates of appropriate influenza and pneumococcal vaccination among adults who receive care at a large multi-specialty group practice in central Massachusetts.

The investigators plan to conduct a non-blinded randomized controlled trial during flu season 2014-2015 (Cycle 1). A total of 20,000 e-portal users and 10,000 non e-portal users who are identified in the Reliant Medical Group (RMG) Electronic Health Record (EHR) as not being up to date on their influenza vaccines will be randomized.

E-portal users will be randomized to receive:

* Arm 1: E-portal message with Interactive Voice Recognition (IVR) call
* Arm 2: E-portal message with no IVR call
* Arm 3: No e-portal message with IVR call OR
* Arm 4: No e-portal message with no IVR call (Control, e-portal users)

Non e-portal users will be randomized to receive either:

* Arm 5: IVR call OR
* Arm 6: no IVR call (Control, non e-portal users)

DETAILED DESCRIPTION:
The study's multifaceted approach will address the gap between current and optimal vaccination rates via patient-, provider- and system-level interventions intended to target local barriers.

Patient-level outreach consisting of education and access information about influenza and pneumococcal vaccines will be delivered through Interactive Voice Recognition (IVR) calls and electronic patient portal messages. The study will have two patient-level outreach cycles. These outreach cycles will address the 2014-2015 flu season (Cycle 1) and the 2015-2016 flu season (Cycle 2).

A non-blinded randomized controlled trial design will be utilized during Cycle 1. A total of 20,000 e-portal users and 10,000 non e-portal users who are identified in the Reliant Medical Group (RMG) Electronic Health Record (EHR) as not being up to date on their influenza vaccines will be randomized. E-portal users will be randomized to receive: (1) E-portal message with Interactive Voice Recognition (IVR) call; (2) E-portal message with no IVR call; (3) No e-portal message with IVR call; or (4) No e-portal message with no IVR call. Non e-portal users will be randomized to receive either (1) IVR call or (2) no IVR call.

In Outreach Cycle 2, investigators will implement a broader outreach effort in which vaccination messages are sent to all e-portal users and IVR messages are sent to 15,000 patients who did not receive vaccinations in the 2014-2015 influenza season. The 15,000 patients receiving IVR calls will be randomly selected.

In an attempt to improve the effectiveness of the intervention in Cycle 2, we will incorporate more detailed information (dates/times/locations on all RMG flu clinics) into both the IVR and e-portal messages. The rate at which e-portal messages can be distributed by RMG will limit the number that can be sent out before the scheduled flu clinics. Patients will therefore be randomly assigned to one of two groups: (A) half of the e-portal users will be sent early messages (approx. 19,000 patients anticipated), while (B) the other half of the e-portal users will not receive early messages. Those in the early message group will receive a message containing flu clinic location, dates, and times. Those in the non-early intervention group will be sent a simplified e-portal message in November 2015 (if they have not already been vaccinated for the 2015-2016 influenza season).

The study team plans to conduct qualitative interviews with 20 patients as well as 10 providers and staff in order to tailor intervention components during Cycle 1.

Provider-level components will include targeted and recurring educational materials for providers and their staff regarding the indications, risks and benefits of influenza and pneumococcal vaccination, and suggesting strategies for overcoming local barriers to vaccination. Beginning in year 2, providers will also receive individualized report cards providing feedback on their immunization rates.

System-level components will include both the capability to capture patient reported vaccinations and automatic updating of EHR vaccination records with pneumococcal and influenza immunizations given at local hospitals and skilled nursing facilities. These system-level components will reduce inappropriate alerts and improve provider confidence in patient records.

The key objectives are:

1. To improve rates of influenza and pneumococcal vaccination in eligible patient populations via:

   1. Patient-level outreach targeted at unvaccinated patients;
   2. Provider- and staff-level educational interventions and system support.
2. To improve the capture of vaccinations administered to Reliant Medical Group (RMG) patients in the community, hospitals and nursing facilities via system-level electronic Health Information Exchange (HIE)

ELIGIBILITY:
Inclusion Criteria:

* RMG Patients 18 years of age or older.
* Overdue for vaccination against influenza and/or not up to date on vaccination for pneumococcal vaccine per RMG EHR data
* No documented allergy to the vaccination in question.

Exclusion Criteria:

* Failure to meet inclusion criteria.
* Patients who have selected the "Do not call" option in the RMG EHR or have an allergy to the influenza and/or pneumococcal vaccination will be excluded from participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30000 (Actual)
Dates: Start 2014-11 (Actual); Primary Completion 2016-06 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sarah L Cutrona, MD, MPH, Principal Investigator — University of Massachusetts, Worcester
Locations (1):
- Reliant Medical Group, Worcester, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wijesundara JG, Ito Fukunaga M, Ogarek J, Barton B, Fisher L, Preusse P, Sundaresan D, Garber L, Mazor KM, Cutrona SL. Electronic Health Record Portal Messages and Interactive Voice Response Calls to Improve Rates of Early Season Influenza Vaccination: Randomized Controlled Trial. J Med Internet Res. 2020 Sep 25;22(9):e16373. doi: 10.2196/16373. PMID 32975529
- [Derived] Cutrona SL, Golden JG, Goff SL, Ogarek J, Barton B, Fisher L, Preusse P, Sundaresan D, Garber L, Mazor KM. Improving Rates of Outpatient Influenza Vaccination Through EHR Portal Messages and Interactive Automated Calls: A Randomized Controlled Trial. J Gen Intern Med. 2018 May;33(5):659-667. doi: 10.1007/s11606-017-4266-9. Epub 2018 Jan 30. PMID 29383550
- [Derived] Cutrona SL, Sreedhara M, Goff SL, Fisher LD, Preusse P, Jackson M, Sundaresan D, Garber LD, Mazor KM. Improving Rates of Influenza Vaccination Through Electronic Health Record Portal Messages, Interactive Voice Recognition Calls and Patient-Enabled Electronic Health Record Updates: Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2016 May 6;5(2):e56. doi: 10.2196/resprot.5478. PMID 27153752

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Cycle 1 Outreach
Groups:
- Arm 1: E-portal Message With IVR Call: Patients identified as e-portal users will receive an e-portal message with Interactive Voice Recognition (IVR) call
  Arm 1: E-portal message with IVR call: Active electronic patient portal users will be randomized to receive an e-portal message and IVR calls. Both methods of outreach will provide patients with educational information about influenza vaccination, notify patients of local flu clinic schedules and elicit patient response to vaccination status and barriers.
Period: Overall Study
Arm/Group | Arm 1: E-portal Message With IVR Call | Arm 2: E-portal Message With no IVR Call | Arm 3: No E-portal Message With IVR Call | Arm 4: No E-portal Message With no IVR Call | Arm 5: IVR Call | Arm 6: No IVR Call
Started | 5000 | 5000 | 5000 | 5000 | 5000 | 5000
Completed | 5000 | 5000 | 5000 | 5000 | 5000 | 5000
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1: E-portal Message With IVR Call | Arm 2: E-portal Message With no IVR Call | Arm 3: No E-portal Message With IVR Call | Arm 4: No E-portal Message With no IVR Call | Arm 5: IVR Call | Arm 6: No IVR Call | Total
Number analyzed (Participants) | 5000 | 5000 | 5000 | 5000 | 5000 | 5000 | 30000
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 4444 | 4416 | 4403 | 4360 | 4320 | 4303 | 26246
  >=65 years | 556 | 584 | 597 | 640 | 680 | 697 | 3754
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3111 | 3179 | 3166 | 3132 | 2497 | 2531 | 17616
  Male | 1889 | 1821 | 1834 | 1868 | 2503 | 2469 | 12384
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 4031 | 4105 | 4022 | 4125 | 3519 | 3554 | 23356
  Black | 150 | 145 | 153 | 113 | 234 | 230 | 1025
  Asian | 252 | 212 | 248 | 211 | 189 | 200 | 1312
  Other | 86 | 72 | 81 | 84 | 138 | 161 | 622
  Missing | 481 | 466 | 496 | 467 | 920 | 855 | 3685

OUTCOME MEASURES:

1. Primary Outcome: Reliant Medical Group (RMG) Patients With Electronic Health Record (EHR) Documentation of Influenza Vaccine Completion for 2014/2015 Season
Description: To determine the impact of our interventions on influenza vaccine completion for the 2014-15 influenza season, we calculated frequencies and performed intention-to-treat bivariate analyses of randomized patients (30,000 patients), assessing whether randomization group was associated vaccine completion. Due to differential rates of vaccination at baseline between portal users and non-users, analyses in these groups were conducted separately. We then performed multivariate logistic regression analyses. We created dummy variables for assignment to the portal message arm (among portal users) and for assignment to the Interactive Voice Recognition (IVR) call arm (among both portal users and, separately, among non-portal users). Including these dummy variables and adjusting for demographic and practice-level covariates, we modeled the odds of receiving an influenza vaccine in the 2014-15 influenza season.
Time Frame: Months 11-16
Population: Using computer-generated random number assignments, we selected 20,000 portal users and 10,000 non portal users (total of 30,000 patients) from the eligible population.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1: E-portal Message With IVR Call | Arm 2: E-portal Message With no IVR Call | Arm 3: No E-portal Message With IVR Call | Arm 4: No E-portal Message With no IVR Call | Arm 5: IVR Call | Arm 6: No IVR Call
Number analyzed (Participants) | 5000 | 5000 | 5000 | 5000 | 5000 | 5000
Participants | 702 | 669 | 642 | 582 | 427 | 430
Statistical Analysis 1: Comparison: Arm 1: E-portal Message With IVR Call vs Arm 4: No E-portal Message With no IVR Call; Test type: Superiority — We calculated frequencies and performed intention-to-treat bivariate analyses. We then performed multivariate logistic regression analyses. With our proposed sample size and using a factorial design, power calculations based on estimates of baseline vaccination rates indicated that 4286 participants per arm would give 80% power to detect a 3% improvement in influenza vaccination rates between groups (α=.05; 2-sided); p = 0.0001, Regression, Logistic — Adjusted for age, sex, race and utilization; Odds Ratio (OR) = 1.30, 95% CI 2-sided [1.15 to 1.47]
Statistical Analysis 2: Comparison: Arm 2: E-portal Message With no IVR Call vs Arm 4: No E-portal Message With no IVR Call; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = .0026, Regression, Logistic; Odds Ratio (OR) = 1.20, 95% CI 2-sided [1.07 to 1.36]
Statistical Analysis 3: Comparison: Arm 3: No E-portal Message With IVR Call vs Arm 4: No E-portal Message With no IVR Call; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = .0206, Regression, Logistic; Odds Ratio (OR) = 1.16, 95% CI 2-sided [1.02 to 1.31]
Statistical Analysis 4: Comparison: Arm 1: E-portal Message With IVR Call vs Arm 2: E-portal Message With no IVR Call; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = .2330, Regression, Logistic; Odds Ratio (OR) = 1.07, 95% CI 2-sided [.96 to 1.21]
Statistical Analysis 5: Comparison: Arm 1: E-portal Message With IVR Call vs Arm 3: No E-portal Message With IVR Call; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = .0579, Regression, Logistic; Odds Ratio, log = 1.12, 95% CI 2-sided [.996 to 1.26]
Statistical Analysis 6: Comparison: Arm 5: IVR Call vs Arm 6: No IVR Call; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = .87, Regression, Logistic; Odds Ratio (OR) = .99, 95% CI 2-sided [.86 to 1.14]

2. Secondary Outcome: Reliant Medical Group (RMG) Patients With Electroinc Health Record (EHR) Documentation of Pneumococcal Vaccine Completion
Description: Using as a denominator those patients identified as being overdue for pneumococcal vaccine at the time of randomization, we calculated frequencies and performed bivariate and multivariate logistic regression analyses, examining the association between randomization group and completion of pneumococcal vaccine. We analyzed portal users and non-portal users separately.
Time Frame: Months 11-16
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1: E-portal Message With IVR Call | Arm 2: E-portal Message With no IVR Call | Arm 3: No E-portal Message With IVR Call | Arm 4: No E-portal Message With no IVR Call | Arm 5: IVR Call | Arm 6: No IVR Call
Number analyzed (Participants) | 1122 | 1164 | 1176 | 1183 | 1580 | 1562
Participants | 153 | 155 | 176 | 178 | 161 | 154
Statistical Analysis 1: Comparison: Arm 1: E-portal Message With IVR Call vs Arm 2: E-portal Message With no IVR Call; Test type: Superiority — Using as a denominator those patients identified as being overdue for pneumococcal vaccine at the time of randomization, we calculated frequencies and performed bivariate and multivariate logistic regression analyses, examining the association between randomization group and completion of pneumococcal vaccine. We analyzed portal users and non-portal users separately; p = .82, Regression, Logistic; Odds Ratio (OR) = 1.03, 95% CI 2-sided [.81 to 1.31]
Statistical Analysis 2: Comparison: Arm 1: E-portal Message With IVR Call vs Arm 3: No E-portal Message With IVR Call; Test type: Superiority — [test comment as in outcome 2, analysis 1]; p = .36, Regression, Logistic; Odds Ratio, log = .90, 95% CI 2-sided [.71 to 1.13]
Statistical Analysis 3: Comparison: Arm 1: E-portal Message With IVR Call vs Arm 4: No E-portal Message With no IVR Call; Test type: Superiority — [test comment as in outcome 2, analysis 1]; p = .33, Regression, Logistic; Odds Ratio (OR) = .89, 95% CI 2-sided [.71 to 1.13]
Statistical Analysis 4: Comparison: Arm 2: E-portal Message With no IVR Call vs Arm 4: No E-portal Message With no IVR Call; Test type: Superiority — [test comment as in outcome 2, analysis 1]; p = .23, Regression, Logistic; Odds Ratio (OR) = .87, 95% CI 2-sided [.69 to 1.09]
Statistical Analysis 5: Comparison: Arm 3: No E-portal Message With IVR Call vs Arm 4: No E-portal Message With no IVR Call; Test type: Superiority — [test comment as in outcome 2, analysis 1]; p = .96, Regression, Logistic; Odds Ratio (OR) = .99, 95% CI 2-sided [.79 to 1.25]
Statistical Analysis 6: Comparison: Arm 5: IVR Call vs Arm 6: No IVR Call; Test type: Superiority — [test comment as in outcome 2, analysis 1]; p = .76, Regression, Logistic; Odds Ratio (OR) = 1.04, 95% CI 2-sided [.82 to 1.31]

3. Other Pre Specified Outcome: Intervention Patients With Self-reported Influenza Vaccinations Documented in Electronic Health Record (EHR)
Description: We calculated the percent of patients who used the portal or IVR to self-report influenza vaccine completion outside of the medical group, measured on April 1, 2015. We used as our denominator all those patients who received portal messages (10,000) and all those who received IVR calls (15,000).
Time Frame: Months 11-16
Measure: Count of Participants; unit: Participants
Groups:
- Portal Self-Report: Patients who received portal questionnaire.
- IVR Self-Report: Patients who received IVR questionnaire.
Arm/Group | Portal Self-Report | IVR Self-Report
Number analyzed (Participants) | 10000 | 15000
Participants | 1527 | 6774

ADVERSE EVENTS:
Description: All-Cause Mortality, Serious, and Other (not including Serious) Adverse Events were not monitored/assessed.
Arm/Group | Arm 1: E-portal Message With IVR Call | Arm 2: E-portal Message With no IVR Call | Arm 3: No E-portal Message With IVR Call | Arm 4: No E-portal Message With no IVR Call | Arm 5: IVR Call | Arm 6: No IVR Call
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
It is possible that our findings are not generalizable to patients in other parts of the country or to those without regular access to primary care.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No